CLINICAL TRIAL: NCT04858347
Title: Clinical and Functional Outcome of the GEMINI SL Fixed Bearing PS Knee Prosthesis in Short-, Mid-, and Longterm Follow-up
Brief Title: Clinical and Functional Outcome of the GEMINI SL Fixed Bearing PS Knee Prosthesis
Status: Recruiting | Type: Observational
Sponsor: Waldemar Link GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: KP11
Record Dates: First submitted 2021-04-14; First posted 2021-04-26 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthrosis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Total knee replacement — Implantation of the GEMINI SL Fixed Bearing PS knee prosthesis. The operation technique of the GEMINI SL Fixed Bearing PS knee prosthesis will be followed.

SUMMARY:
This is a prospective, multicenter, observational study with a planned follow-up period of 10 years to confirm the safety and performance of the GEMINI SL Fixed Bearing PS knee prosthesis in longterm follow-up under routine conditions. Primary outcome of the study is the 10-year survival rate of the GEMINI SL Fixed Bearing PS knee prosthesis with revision for any reason as the endpoint.

DETAILED DESCRIPTION:
The GEMINI SL Fixed Bearing PS knee prosthesis combines clinical proven design features with state-of-the-art-technology in order to achieve a high standard clinical performance, surgical efficiency and safety. Currently, no mid- and longterm clinical data are available for the GEMINI SL Fixed Bearing PS knee prosthesis. Therefore, the study is designed to generate clinical data of the GEMINI SL Fixed Bearing PS knee prosthesis in the 10-year follow-up under routine condition.

ELIGIBILITY:
Inclusion Criteria:

* Signed patient informed consent
* Implantation of a GEMINI SL Fixed Bearing PS knee prosthesis
* Age between 18 and 80 years

Exclusion Criteria:

* Body Mass Index (BMI) > 40 kg/m²
* Foreseeable life expectancy under 5 years
* Comorbidities and known medical circumstances which would affect the clinical or functional outcome after implantation of the knee prosthesis (e.g. neurological or musculoskeletal diseases) at the time of implantation
* Patient who is mentally not able to understand the study and the study conduct
* Patients who will be foreseeable non-compliant to the planned routine interventions and study related follow-ups
* Prisoner
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are scheduled for an implantation of the GEMINI SL Fixed Bearing PS knee prosthesis are potential study participants. The decision about the surgical treatment and the use of the GEMINI SL Fixed Bearing PS knee prosthesis is made by the treating surgeons and depends on Link Gemini SL Fixed Bearing PS _ Colombia Version 1.0 vom 24.08.2018 Seite 12 von 19 the clinical findings of the patient. The potential study participation is independent from the therapy decision.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2034-10 (Estimated); Study Completion 2035-10 (Estimated)

PRIMARY OUTCOMES:
10-year survival rate of the Gemini SL Fixed Bearing PS knee prothesis | 10 years
  Primary outcome of the study is the 10-year survival rate of the Gemini SL Fixed Bearing PS knee prosthesis with revision for any reason as the endpoint. Revisions are defined as removal, exchange or adding of any implant components. The definition does not include subsequent implantations or exchange of the patella component or the polyethylene plateau. Survival rate will be calculated according to the method of Kaplan-Meier.

SECONDARY OUTCOMES:
Survival rate of the GEMINI SL Fixed Bearing PS knee prosthesis | after 6 months, 1,3 and 5 years
  Survival rate of the GEMINI SL Fixed Bearing PS knee prosthesis after 6 months, 1, 3 and 5 years
Change in functional and clinical outcome (KOOS) | preoperative examination to postoperative examinations after 6 months, 1, 3, 5 and 10 years
  Evaluation of the change in functional and clinical outcome from preoperative to 6 months, 1, 3, 5 and 10 years postoperative, measured by the Knee injury and Osteoarthritis Outcome Score (KOOS). The KOOS is a reliable and validated knee-specific patient-administered outcome instrument. The previous week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 (best result) to 4 (worst result). The KOOS consists of 5 sub-scales: Pain, Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and Hip/Knee related Quality of life (QoL). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Change in functional and clinical outcome (KSS) | preoperative examination to postoperative examinations after 6 months, 1, 3, 5 and 10 years
  Evaluation of the change in functional and clinical outcome from preoperative to 6 months, 1, 3, 5 and 10 years postoperative, measured by the Knee Society Score (KSS). The KSS is a frequently used, reliable and validated score in the assessment of a subject's knee pain and functional knee capacity. It comprises two arms, the functional ability and the clinical examination score, each ranging from 0 points (worst result) to 100 points (best result).
Complications rate | Intraoperative examinations to 10-year follow-up examination
  Complications related to implantation of the GEMINI SL Fixed Bearing PS knee prosthesis (infections, dislocations, migrations, aseptic loosenings, periprosthetic fractures, intra-operative fractures, implant fractures, soft tissue fractures, joint instability etc.) will be recorded at all follow-up examinations.
Subsequent surgical interventions | postoperative examinations up to 10-year follow-up examination
  All subsequent surgical interventions at the operated knee (exchange of the polyethylene plateau, additional implantation/exchange of the patella component, soft-tissue balancing, debridement etc) will be recorded at all follow-up examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Cesar Palacio Villegas, Dr., Principal Investigator — Centro Medico Imbanaco Sede Principal
Locations (1):
- Centro Medico Imbanaco Sede Principal, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No